CLINICAL TRIAL: NCT01645098
Title: Sedation During Muscle Biopsy in Patients With Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB11-00532
Record Dates: First submitted 2012-06-08; First posted 2012-07-20 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine 1 mcg/kg (Experimental): Patients receive a loading dose of dexmedetomidine 1 mcg/kg followed by a continuous infusion of 1 mcg/kg/hr.
  Interventions: Drug: Ketamine; Drug: Dexmedetomidine
- Dexmedetomidine 0.5 mcg/kg (Experimental): Patients receive a loading dose of dexmedetomidine 0.5 mcg/kg followed by a continuous infusion of 0.5 mcg/kg/hr.
  Interventions: Drug: Ketamine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ketamine — 1 mg/kg IV, additional doses of 0.5 mg/kg as needed
Drug: Dexmedetomidine — 0.5 mcg/kg/hr IV

SUMMARY:
This is an interventional study on Duchenne muscular dystrophy patients who will be receiving sedation for a muscle biopsy as part of another study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a muscle biopsy for IRB11-00203.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-08; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine 1 mcg/kg | Dexmedetomidine 0.5 mcg/kg
Started | 24 | 29
Completed | 24 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine 1 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Total
Number analyzed (Participants) | 24 | 29 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (1.4) | 8.9 (1.9) | 9.4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 29 | 53

OUTCOME MEASURES:

1. Primary Outcome: Time to Sedation Score of 3-4
Description: The depth of sedation was judged using the University of Michigan Sedation Scale (UMSS). The score ranges from zero, awake and alert, to four, unarousable. A score of three, deeply sedated, or more was considered to be an appropriate level of sedation for the procedure.
Time Frame: Immediately prior to incision
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dexmedetomidine 1 mcg/kg | Dexmedetomidine 0.5 mcg/kg
Number analyzed (Participants) | 24 | 29
minutes | 3.7 (2.3) | 2.8 (1.6)

2. Secondary Outcome: Heart Rate Change After Dexmedetomidine Loading Dose
Description: Difference in heart rate from baseline to immediately following infusion of dexmedetomidine loading dose.
Time Frame: Baseline to immediately post dexmedetomidine infusion.
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Dexmedetomidine 1 mcg/kg | Dexmedetomidine 0.5 mcg/kg
Number analyzed (Participants) | 24 | 29
BPM | -13 (13) | -5 (10)

3. Secondary Outcome: Mean Arterial Pressure (MAP) Change After Dexmedetomidine Loading Dose
Description: Change in MAP from baseline measurement to immediately post dexmedetomidine infusion measured via blood pressure cuff.
Time Frame: Baseline to immediately post dexmedetomidine infusion.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine 1 mcg/kg | Dexmedetomidine 0.5 mcg/kg
Number analyzed (Participants) | 24 | 29
mmHg | 9 (10) | 5 (8)

4. Secondary Outcome: Oxygen Saturation Change After Dexmedetomidine Loading Dose
Description: Change in oxygen saturation from baseline measurement to immediately post dexmedetomidine infusion.
Time Frame: Baseline to immediately post dexmedetomidine infusion.
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | Dexmedetomidine 1 mcg/kg | Dexmedetomidine 0.5 mcg/kg
Number analyzed (Participants) | 24 | 29
percentage of oxygen | -0.3 (1.2) | 0.4 (0.7)

5. Secondary Outcome: EtCO2 Change After Dexmedetomidine Loading Dose
Description: Change in end-tidal carbon dioxide from baseline measurement to immediately post dexmedetomidine infusion.
Time Frame: Baseline to immediately post dexmedetomidine infusion.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine 1 mcg/kg | Dexmedetomidine 0.5 mcg/kg
Number analyzed (Participants) | 24 | 29
mmHg | 1 (5) | 2 (6)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine 1 mcg/kg | Dexmedetomidine 0.5 mcg/kg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/29
Other Adverse Events (participants affected / at risk) | 0/24 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes